CLINICAL TRIAL: NCT06356597
Title: Division of Gastroenterology and Hepatology,Renji Hospital, School of Medicine, Shanghai Jiao Tong University
Brief Title: Tislelizumab With Fruquintinib, Metronidazole, in Mismatch Repair-proficient or Microsatellite Stability, Advanced Colorectal Cancer: a Multicenter, Single Arm, Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jing-yuan Fang, MD, Ph. D (Other)
Responsible Party: Sponsor-Investigator, Jing-yuan Fang, MD, Ph. D, Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-004-A
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; HMPL-013; Metronidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab with Fruquintinib, Metronidazole (Experimental)
  Interventions: Drug: Tislelizumab with Fruquintinib, Metronidazole

INTERVENTIONS:
Drug: Tislelizumab with Fruquintinib, Metronidazole — Metronidazole tablets: One administration cycle is every 6 weeks, and metronidazole tablets are given orally on the 1st to 7th day of each cycle. The medication method is two tablets three times one day.
  Teralizumab: Every 3 weeks is a dosing cycle, with 200mg of Teralizumab administered intravenously on the first day of each cycle.

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of Tislelizumab with Fruquintinib, Metronidazole treatment in MSS/MSI-L advanced colorectal cancer patients with high abundance of Fusobacterium nucleatum in a single arm Phase II clinical.

ELIGIBILITY:
Inclusion Criteria:

1. No gender limit, age ≥ 18 years old and ≤ 80 years old;
2. Colorectal cancer (AJCC stage IV) diagnosed by histological or cytological biopsy as metastatic or unresectable, with immunohistochemical or genetic testing indicating MSS or MSH-L type;
3. Treatment requires third line or above, has previously received standard first and second line treatment, and the disease has progressed after treatment;
4. Before accepting tirelizumab, qPCR should be used to detect the Fn deltaCT value ≥ -22.24 in fecal samples;
5. ECOG score: 0-1 points;
6. Baseline blood routine and biochemical indicators meet the following criteria (no blood transfusion or use of colony stimulating factors 2 weeks prior to screening) Blood routine: hemoglobin ≥ 90g/L, absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet ≥ 100 × 109/L Liver function: ALT and AST ≤ 2.5 x ULN, serum total bilirubin ≤ 1.5 x ULN (if there is liver metastasis, ALT and AST ≤ 5 x ULN, serum total bilirubin ≤ 3 x ULN), serum albumin ≥ 30g/L Renal function: serum creatinine ≤ 1.5 x upper limit of normal (ULN), or creatinine clearance rate ≥ 50 mL/min (calculated according to Cockcroft Gault formula).
7. Those who voluntarily participate in the trial and sign an informed consent form.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Chronic intestinal diseases (such as Crohn's disease, ulcerative colitis, etc.), infectious intestinal diseases during the screening period, and intestinal obstruction during the screening period;
3. Subjects with poor control of hypertension (systolic blood pressure>150 mmHg and/or diastolic blood pressure>100 mmHg) and a history of hypertensive crisis or hypertensive brain disease;
4. Severe liver and kidney function or heart dysfunction;
5. Patients who use antibiotics for more than 5 days within one month prior to immunotherapy;
6. Patients with known brain or meningeal metastases, regardless of whether they have received treatment, are not eligible for inclusion in this trial.
7. Individuals with contraindications to the use of metronidazole medication;
8. Those who are unwilling to participate in the trial or sign informed consent forms;
9. The researchers believe that there are any situations that are not suitable for selection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2027-12-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 3 months and 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Ninth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Jiang SS, Xie YL, Xiao XY, Kang ZR, Lin XL, Zhang L, Li CS, Qian Y, Xu PP, Leng XX, Wang LW, Tu SP, Zhong M, Zhao G, Chen JX, Wang Z, Liu Q, Hong J, Chen HY, Chen YX, Fang JY. Fusobacterium nucleatum-derived succinic acid induces tumor resistance to immunotherapy in colorectal cancer. Cell Host Microbe. 2023 May 10;31(5):781-797.e9. doi: 10.1016/j.chom.2023.04.010. Epub 2023 May 1. PMID 37130518